CLINICAL TRIAL: NCT07366307
Title: Management of Indwelling Labor Epidural Catheters and Pain During Cesarean Delivery: a Prospective Single-center Patient-reported Outcome Study
Brief Title: Management of Indwelling Labor Epidural Catheters for Cesarean Delivery
Status: Not yet recruiting | Type: Observational
Sponsor: Baylor Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: 025-604
Record Dates: First submitted 2026-01-02; First posted 2026-01-26 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2025-12

CONDITIONS: Intraoperative Pain
Keywords: cesarean section; pain; labor epidural catheter; top up
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cesarean delivery patients: Patients who had an indwelling labor epidural catheter and subsequently underwent cesarean delivery.

SUMMARY:
This is a prospective observational study that will survey patients who had an indwelling labor epidural catheter and subsequently underwent cesarean delivery. We hypothesize that patients who had removal of indwelling labor epidural catheters and had a new neuraxial anesthetic technique attempted will have a lower incidence of self-reported pain during cesarean delivery compared to patients who had top up of their indwelling labor epidural catheters.

ELIGIBILITY:
Inclusion Criteria:

* ages 18-50 years
* had cesarean delivery at Baylor Scott & White Medical Center from January 1, 2026 through December 31, 2026
* Fluent in the English language (our catastrophizing survey is validated in English language only)
* Can provide their own consent
* Identifies as Black or African American only, Hispanic, or White or Caucasian only
* had administration of local anesthetic through indwelling labor epidural or removal of indwelling labor epidural followed by single injection spinal or combined spinal epidural

Exclusion Criteria:

* less than 18 years old, older than 50 years old
* had cesarean delivery at Baylor Scott & White Medical Center before January 1, 2026 or after December 31, 2026
* Employee of Baylor Scott & White Health labor and delivery unit
* Student of a school that performs clinical rotations at Baylor Scott & White Medical Center-Temple
* Incarcerated at the time of study enrollment
* Underwent scheduled cesarean hysterectomy
* Underwent cesarean delivery with general anesthesia as either the primary anesthetic technique or had conversion to general anesthesia because of failure of neuraxial anesthesia
* Admitted to the intensive care unit immediately following cesarean delivery
* Did not have intrathecal morphine or intrathecal fentanyl if receiving spinal anesthesia
* Had anesthesia for an attempted external cephalic version within 24 hours of cesarean delivery

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Patients will be identified as potential study participants if they have a cesarean delivery at Baylor Scott & White Medical Center-Temple from January 1, 2026 through December 31, 2025.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Pain during cesarean delivery | Patients will be asked this question once 24-72 hours after their cesarean delivery.
  Patients will answer "yes" or "no" to whether they experienced pain during their cesarean delivery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael P Hofkamp, M.D., Principal Investigator — Baylor Scott & White Medical Center-Temple

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Litman J, Bates R, Lindheim SR, Sharpe EE, Ehrig JC, Hofkamp MP. Patient and clinical characteristics associated with pain during cesarean delivery: a prospective single-center patient-reported outcome study. Int J Obstet Anesth. 2025 Feb;61:104324. doi: 10.1016/j.ijoa.2024.104324. Epub 2025 Jan 10. PMID 39827661

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2025-12-16): https://cdn.clinicaltrials.gov/large-docs/07/NCT07366307/Prot_SAP_000.pdf
  • Informed Consent Form (2025-12-15): https://cdn.clinicaltrials.gov/large-docs/07/NCT07366307/ICF_001.pdf